CLINICAL TRIAL: NCT02311985
Title: Point-of-care Versus Standard Coagulation Tests Versus Restrictive Strategy to Guide Transfusion in Chronic Liver Failure Patients Requiring Central Venous Line: Prospective Randomized Trial
Brief Title: Comparison of Three Transfusion Strategies for Central Venous Catheterization in Cirrhotics: A Randomized Clinical Trial
Acronym: POCKET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low inclusion rate
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Leonardo Lima Rocha, MD, Adult Critical Care Medicine Attending Physician, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2048-14
Record Dates: First submitted 2014-12-03; First posted 2014-12-09 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; Blood coagulation; Thromboelastography; Blood transfusion; Catheterization, central venous
MeSH Terms: conditions — Liver Cirrhosis; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Coagulogram-based protocol (Active Comparator): Arm based on standard coagulation tests protocol to guide blood transfusion before central venous catheterization. The possible components to be used include fresh frozen plasma, platelets (random or aphaeresis) and or cryoprecipitate.
  Interventions: Other: Coagulogram-based protocol
- Thromboelastometry-based protocol (Experimental): Arm based on rotational thromboelastometry (ROTEM(R)) protocol to guide blood transfusion before central venous catheterization. The possible components to be used include fresh frozen plasma, platelets (random or aphaeresis) and or cryoprecipitate.
  Interventions: Other: Thromboelastometry-based protocol
- Restrictive strategy (Experimental): Arm based on a restrictive protocol strategy based on INR/PT and platelets count. The possible components to be used include fresh frozen plasma and/or platelets (random or aphaeresis).
  Interventions: Other: Restrictive strategy

INTERVENTIONS:
Other: Coagulogram-based protocol — The interventions for this protocol include transfusion of fresh frozen plasma, platelets (random or aphaeresis) and/or cryoprecipitate, based on international normalised ratio (INR), partial thromboplastin time (PTT), platelet count and/or fibrinogen. If INR >1.5 or PTT >50 sec., fresh frozen plasma is administered (dose: 10 mL/Kg); and/or platelets <50,000/microliter, random or aphaeresis platelets are administered (01 unit/Kg or 01 aphaeresis); and/or fibrinogen <150 mg/dL, cryoprecipitate is administered (dose: 01 unit/Kg).
  Arms: Coagulogram-based protocol
Other: Thromboelastometry-based protocol — The interventions for this protocol include transfusion of fresh frozen plasma, platelets (random or aphaeresis) and/or cryoprecipitate, based on rotational thromboelastometry (ROTEM(R)). If CTex <80 sec. and A10ex >40 mm, then no blood transfusion is performed; when CTex >80s, then fresh frozen plasma is administered (dose: 10 mL/Kg); and/or A10ex <40 mm or A10fib >10 mm, random or aphaeresis platelets are administered (01 unit/Kg or 01 aphaeresis); and/or A10ex <40 mm or A10fib <10 mm, cryoprecipitate is administered (dose: 01 unit/Kg).
  Arms: Thromboelastometry-based protocol
Other: Restrictive strategy — The interventions for this protocol include transfusion of fresh frozen plasma and/or platelets (random or aphaeresis), based on INR and platelet count. If INR >5, fresh frozen plasma is administered (dose: 10 mL/Kg); and/or platelets <25,000/microliter, random or aphaeresis platelets are administered (01 unit/Kg or 01 aphaeresis).
  Arms: Restrictive strategy

SUMMARY:
The aim of this study is to compare three different blood transfusion strategies for coagulopathy correction before central venous catheterization in patients with chronic liver failure (cirrhosis and/or chronic liver graft dysfunction) admitted in intensive care unit.

DETAILED DESCRIPTION:
Central venous catheterization is a ubiquitous procedure in intensive care units and is mainly used for drug administration, hemodynamic monitoring and hemodialysis. Only in US more than five million catheters are inserted annually. One of the main complications associated to central venous lines are the mechanical ones, i.e. arterial puncture, bleeding and hematoma formation, which varies between 5% and 19%. The use of real-time ultrasonography to accomplish central venous catheterization was associated to a drastic reduction in complication rates, and when performed by trained personnel, some series show complications rates <1%, even in patients with coagulopathy.

Patients presenting with chronic liver failure has a complex coagulation system balance, resulting from reduction in the majority of procoagulant and anticoagulant factors, opposed by preservation of thrombin generation. Thus, these patients are prone to develop hemorrhagic and thrombotic phenomena. The coagulation of cirrhotic patients have been classically evaluated by standard coagulation tests. Nevertheless, these tests present important limitations, as evaluation of plasmatic component only, and do not predict bleeding risk. The thromboelastometry is a point-of-care real-time coagulation system evaluation with the advantage of evaluating the cellular and plasmatic components of the coagulation and present a more comprehensive evaluation of blood coagulation, specially in cirrhotics. This technology is associated with reduced costs in diverse clinical settings.

In clinical practice, approximately 90% of physicians empirically transfuse blood components to cirrhotic patients before invasive procedures. This practice is associated to increased risks related to blood transfusion per se, e.g. blood borne infections, immunologic and non-immunologic adverse reactions, to cite some. Several randomized clinical trials have shown that restrictive blood transfusion strategies are associated to better outcomes, including mortality.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver failure (cirrhosis or chronic graft dysfunction) from any cause and medical indication of central venous line placement

Exclusion Criteria:

* Acute liver failure or
* Use of therapeutic doses of oral or parenteral anticoagulants (unfractionated heparin or low molecular weight heparin or oral anticoagulants) or
* Use of oral or parenteral platelet aggregation inhibitors or
* Patients with von Willebrand syndrome or
* Over-the-guidewire central venous catheter changing
* Patients previously included in this study protocol during the same hospital stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients submitted to blood components transfusion - i.e. fresh frozen plasma, platelets and/or cryoprecipitate - before central venous catheterization | Day of randomization

SECONDARY OUTCOMES:
Incidence of hemorrhagic complications associated to central venous catheterization procedure | Day 1
Incidence of acute immunologic and non-immunologic adverse effects of blood transfusion | Day 1
Costs assessments (laboratory and blood transfusion) between the three strategies | Day 1
Length of stay in ICU | Up to 90 days
Length of stay in hospital | Up to 180 days
Mortality rate | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Silva, MD, PhD, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Background] Tercan F, Ozkan U, Oguzkurt L. US-guided placement of central vein catheters in patients with disorders of hemostasis. Eur J Radiol. 2008 Feb;65(2):253-6. doi: 10.1016/j.ejrad.2007.04.002. Epub 2007 May 4. PMID 17482407
- [Background] Tripodi A, Mannucci PM. The coagulopathy of chronic liver disease. N Engl J Med. 2011 Jul 14;365(2):147-56. doi: 10.1056/NEJMra1011170. No abstract available. PMID 21751907
- [Background] Stravitz RT. Potential applications of thromboelastography in patients with acute and chronic liver disease. Gastroenterol Hepatol (N Y). 2012 Aug;8(8):513-20. PMID 23293564
- [Background] Segal JB, Dzik WH; Transfusion Medicine/Hemostasis Clinical Trials Network. Paucity of studies to support that abnormal coagulation test results predict bleeding in the setting of invasive procedures: an evidence-based review. Transfusion. 2005 Sep;45(9):1413-25. doi: 10.1111/j.1537-2995.2005.00546.x. PMID 16131373
- [Background] Schochl H, Nienaber U, Maegele M, Hochleitner G, Primavesi F, Steitz B, Arndt C, Hanke A, Voelckel W, Solomon C. Transfusion in trauma: thromboelastometry-guided coagulation factor concentrate-based therapy versus standard fresh frozen plasma-based therapy. Crit Care. 2011;15(2):R83. doi: 10.1186/cc10078. Epub 2011 Mar 4. PMID 21375741
- [Background] Watson DM, Stanworth SJ, Wyncoll D, McAuley DF, Perkins GD, Young D, Biggin KJ, Walsh TS. A national clinical scenario-based survey of clinicians' attitudes towards fresh frozen plasma transfusion for critically ill patients. Transfus Med. 2011 Apr;21(2):124-9. doi: 10.1111/j.1365-3148.2010.01049.x. Epub 2010 Nov 10. PMID 21062383
- [Background] Stanworth SJ, Walsh TS, Prescott RJ, Lee RJ, Watson DM, Wyncoll D; Intensive Care Study of Coagulopathy (ISOC) investigators. A national study of plasma use in critical care: clinical indications, dose and effect on prothrombin time. Crit Care. 2011;15(2):R108. doi: 10.1186/cc10129. Epub 2011 Apr 5. PMID 21466676
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381
- [Background] Carson JL, Terrin ML, Noveck H, Sanders DW, Chaitman BR, Rhoads GG, Nemo G, Dragert K, Beaupre L, Hildebrand K, Macaulay W, Lewis C, Cook DR, Dobbin G, Zakriya KJ, Apple FS, Horney RA, Magaziner J; FOCUS Investigators. Liberal or restrictive transfusion in high-risk patients after hip surgery. N Engl J Med. 2011 Dec 29;365(26):2453-62. doi: 10.1056/NEJMoa1012452. Epub 2011 Dec 14. PMID 22168590
- [Background] Villanueva C, Colomo A, Bosch A, Concepcion M, Hernandez-Gea V, Aracil C, Graupera I, Poca M, Alvarez-Urturi C, Gordillo J, Guarner-Argente C, Santalo M, Muniz E, Guarner C. Transfusion strategies for acute upper gastrointestinal bleeding. N Engl J Med. 2013 Jan 3;368(1):11-21. doi: 10.1056/NEJMoa1211801. PMID 23281973
- [Derived] Rocha LL, Neto AS, Pessoa CMS, Almeida MD, Juffermans NP, Crochemore T, Rodrigues RR, Filho RR, de Freitas Chaves RC, Cavalheiro AM, Prado RR, Assuncao MSC, Guardia BD, Silva E, Correa TD. Comparison of three transfusion protocols prior to central venous catheterization in patients with cirrhosis: A randomized controlled trial. J Thromb Haemost. 2020 Mar;18(3):560-570. doi: 10.1111/jth.14672. Epub 2019 Dec 2. PMID 31667992
- [Derived] Rocha LL, Pessoa CM, Neto AS, do Prado RR, Silva E, de Almeida MD, Correa TD; POCKET Trial Investigators. Thromboelastometry versus standard coagulation tests versus restrictive protocol to guide blood transfusion prior to central venous catheterization in cirrhosis: study protocol for a randomized controlled trial. Trials. 2017 Feb 27;18(1):85. doi: 10.1186/s13063-017-1835-5. PMID 28241780